CLINICAL TRIAL: NCT02715557
Title: Arise: An Online Relapse Prevention Tool for Adolescent Substance Abusers
Acronym: ARISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HHSN27120140075C
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Access to the relapse prevention program (Experimental): The participants will receive access to the relapse prevention program throughout the entire 6-week trial period.
  Interventions: Behavioral: Relapse prevention program
- TAU (Experimental): The participants will receive treatment as usual (TAU) for 6-weeks, and will receive access to the relapse prevention program after the completion of the 6 month follow-up.
  Interventions: Behavioral: Relapse prevention program

INTERVENTIONS:
Behavioral: Relapse prevention program — The relapse prevention program is an innovative computer-based coping skills educational program for adolescent substance abuse treatment completers.

SUMMARY:
In Phase I of this SBIR project, 3C Institute (3C) developed a working prototype of an innovative computer-based coping skills educational program for adolescent substance abuse treatment completers. For Phase I, 3C developed and tested two customizable intelligent educational modules to teach coping skills in order to help adolescents avoid relapse, along with a brief instructional game for each segment. The Phase I prototype also included an online Parent Guide to inform parents about the uses and benefits of the product. Phase I R&D provided strong support for the quality and value of the prototype as well as the viability of the proposed educational package and its promise for preventing substance abuse relapse with adolescents. Phase I results supported excellent quality of the product through high ratings of quality, appeal, and value. High feasibility and usability was also demonstrated through high ratings for ease of use, usability, and potential effectiveness.

The goal of this Phase II SBIR project is to modify and expand the relapse prevention program developed in Phase I in response to customer feedback and to evaluate the efficacy of the full program with an RCT pilot clinical study. This product will be an adaptable software program for aftercare therapy. In Phase II, the investigators will build on the Phase I findings to modify and extend the existing content and develop the full program, which will include: an introductory module as well as interactive lessons and skill-building games for five coping skills modules. The Phase II product will also include a HelpCenter to support sustained, quality use of the product during commercialization.

DETAILED DESCRIPTION:
Purpose:

In Phase I of this SBIR project, 3C Institute (3C) developed a working prototype of an innovative computer-based coping skills educational program for adolescent substance abuse treatment completers. For Phase I, 3C developed and tested two customizable intelligent educational modules to teach coping skills in order to help adolescents avoid relapse, along with a brief instructional game for each segment. The Phase I prototype also included an online Parent Guide to inform parents about the uses and benefits of the product. Phase I R&D provided strong support for the quality and value of the prototype as well as the viability of the proposed educational package and its promise for preventing substance abuse relapse with adolescents. Phase I results supported excellent quality of the product through high ratings of quality, appeal, and value. High feasibility and usability was also demonstrated through high ratings for ease of use, usability, and potential effectiveness.

The goal of this Phase II SBIR project is to modify and expand the relapse prevention program developed in Phase I in response to customer feedback and to evaluate the efficacy of the full program with an RCT pilot clinical study. This product will be an adaptable software program for aftercare therapy. In Phase II, the investigators will build on the Phase I findings to modify and extend the existing content and develop the full program, which will include: an introductory module as well as interactive lessons and skill-building games for five coping skills modules. The Phase II product will also include a HelpCenter to support sustained, quality use of the product during commercialization.

Research Design:

Throughout development and iterative usability testing, the project consultants, experts in the field of adolescent substance abuse treatment and prevention, will review and interact with the relapse prevention program, and results will be used to modify and finalize the user interface and navigation to maximize usability prior to pilot testing with adolescents. Once all revisions and additions have been completed and integrated into the fully functioning product, the investigators will conduct an RCT pilot clinical study with up to 125 adolescents aged 13 - 19 years in substance abuse recovery to evaluate the benefits and effectiveness of the program. The investigators will use a rolling enrollment randomized control design in which adolescents will be randomly assigned to one of two conditions: (a) Group A, in which participants will receive access to the relapse prevention program throughout the entire 6-week trial period, or (b) Group B, in which participants will receive treatment as usual (TAU) for 6-weeks, and will receive access to the relapse prevention program following the completion of all data collection. Over the trial, the following outcome areas will be assessed: substance use and cravings, substance abuse recovery and relapse knowledge, perceived benefits of substance use, coping behaviors and coping, stage of change, and treatment as usual description. The investigators will also assess usability and acceptability of the program and gather information on adverse events/serious adverse events that occur during interaction with the program.

Hypotheses:

Based on Phase I findings and 3C's experience developing similar products, the investigators expect high user ratings on the relapse prevention program, and anticipate greater improvement in outcomes across all areas for adolescents who received access to the relapse prevention program (Group A) compared with those who did not (Group B), providing evidence for the promise of this new educational program for generating beneficial substance use abstinence outcomes. The investigators do not expect participation in the program to be associated with any negative outcomes. The investigators expect Phase II findings to demonstrate greater sobriety maintenance for adolescents with access to the relapse prevention program compared to those in typical aftercare activities.

Length of Study:

The investigators anticipate the pilot phase of this study, including recruitment, conducting the pilot RCT, and collecting follow-up data to last 17 months.

Confidentiality:

Due to the sensitive nature of this study, the investigators have obtained a Certificate of Confidentiality from NIDA. The Certificate number is CC-DA-16-061, and is valid from 9/17/2014 - 9/17/2018.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 - 19 years at time of enrollment
* Met DSM-5 criteria for any substance use disorder preceding primary treatment
* Completed substance abuse treatment within 90 days prior to the start of the trial
* Proficient in reading and writing English
* Access to a computer or tablet with high-speed internet

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in frequency of substance. | (1) within one week prior to the 6-week trial (baseline), (2) within one week of the end of the trial (end-point), and (3) 3 or 6 months after completion of the trial period (follow-up)
  As directed by the contract, the investigators will use the NIDA Common Data Element Timeline Follow-Back measure (TLFB; Sobell & Sobell, 1992) for self-report. Adolescents will complete the TLFB reporting past 30 day use. Adolescents will be presented with a calendar showing the previous 30 days and will be asked to indicate whether or not they used substances each day. For days in which either alcohol or tobacco use is indicated, adolescents will be asked to report the quantity used. The investigators will also measure substance use with a toxicology report. The participant will submit an oral swab for toxicology screening directly to the third-party laboratory, LabCorp, which will evaluate oral swabs for 10 different substances. After the results have been read, the toxicology analyses will be emailed to study staff with the de-identified study number.

SECONDARY OUTCOMES:
Change from baseline in coping behaviors. | (1) within one week prior to the 6-week trial (baseline), (2) within one week of the end of the trial (end-point), and (3) 3 or 6 months after completion of the trial period (follow-up)
  Participants will complete the Coping Behaviors Inventory: (CBI; Litman, Stapleton, Oppenheim, & Peleg, 1983; additional items added by Dr. Sanchez) to report how often they have used a variety of coping skills using this 44-item self-report measure designed to assess coping skills among adolescents with a history of alcohol and other drug abuse.
Change from baseline in knowledge of substance abuse recovery and relapse. | (1) within one week prior to the 6-week trial (baseline), (2) within one week of the end of the trial (end-point), and (3) 3 or 6 months after completion of the trial period (follow-up)
  This investigator-created 20 item measure assesses knowledge of substance abuse relapse risk and prevention and is based on the substance abuse recovery and relapse literature and established measures that have been used to assess substance use.
Change from baseline in perceived benefits of substance use. | (1) within one week prior to the 6-week trial (baseline), (2) within one week of the end of the trial (end-point), and (3) 3 or 6 months after completion of the trial period (follow-up)
  In this 5-item measure, adolescents report the extent to which they believe there are favorable aspects to substance use.
Change from baseline in self-efficacy to avoid substance use. | (1) within one week prior to the 6-week trial (baseline), (2) within one week of the end of the trial (end-point), and (3) 3 or 6 months after completion of the trial period (follow-up)
  Adolescents will complete the Drug Avoidance Self-Efficacy Scale (Martin, G.W., Wilkinson, D.A., & Poulos, C.X., 1995) a 16-item measure of self-efficacy to avoid substance use.
Change from baseline in Readiness of Change. | (1) within one week prior to the 6-week trial (baseline), (2) within one week of the end of the trial (end-point), and (3) 3 or 6 months after completion of the trial period (follow-up)
  Adolescents will complete the 12-item Readiness to Change Questionnaire (Heather, N., & Honekopp, J., 2008) indicating their current stage of change in substance use abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Scrimgeour, Ph.D., Principal Investigator — 3-C Institute for Social Development, dba 3C Institute; Melissa E DeRosier, PhD, Principal Investigator — 3-C Institute for Social Development, dba 3C Institute
Locations (1):
- 3-C Institute for Social Development, dba 3C Institute, Durham, North Carolina, United States